CLINICAL TRIAL: NCT03026218
Title: Group and Mobile Care for Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Sarah Crimmins, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00071275
Record Dates: First submitted 2017-01-11; First posted 2017-01-20 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group and Glucose Mama (Experimental): Enrolled subjects with have GlucoseMama application and group care.
  Interventions: Other: GlucoseMama application with blood sugar monitoring and carb monitoring.; Other: Group prenatal care for GDM.
- Group and No Glucose Mama (Placebo Comparator): Enrolled participants will be enrolled in group care but will not have access to GlucoseMama application.
  Interventions: Other: Group prenatal care for GDM.
- Traditional and glucoseMama (Experimental): Enrolled subjects will have traditional care and glucoseMama
  Interventions: Other: GlucoseMama application with blood sugar monitoring and carb monitoring.
- Traditional and no GlucoseMama (No Intervention): enrolled subjects will not have access to group care or GlucoseMama.

INTERVENTIONS:
Other: GlucoseMama application with blood sugar monitoring and carb monitoring. — We will use the Glucosemama application to review glucose and carb logs on a weekly basis. This will be reviewed with the patient in order to adjust dietary and medicals.
  Arms: Group and Glucose Mama; Traditional and glucoseMama
Other: Group prenatal care for GDM. — group prenatal care is a group based intervention where individuals with GDM will meet together to learn about pregnancy and diabetes.
  Arms: Group and Glucose Mama; Group and No Glucose Mama

SUMMARY:
A critical variation in the provision of prenatal care to women with GDM is the need to keep patients engaged with their care between visits by tracking glucose levels using finger sticks and making dietary and other lifestyle modifications to keep these levels at or close to normal. Multiple studies have demonstrated that the use of mobile devices can improve medical outcomes. In order to keep patients engaged between appointments and improve self-care/lifestyle, we will study the use of a glucose monitoring system with nutrition therapy called GlucoseMama(GM). GM is a mobile app on the iOS system that individuals with GDM will use to tract blood sugars and number of carbs consumed. In addition, it will give the user positive feedback and rewards for using the system. This model of group care with mobile phone monitoring and reminders for women with GDM has not been previously studied. A randomized control trial is purposed to determine if this approach improves patient care. The investigators hypothesize that group prenatal care along with inter-session mobile therapy will increase dietary compliance and therefore reduce the number of individuals requiring pharmacologic therapy and improve neonatal outcomes during pregnancy. Group prenatal care (GPC) will provide a community foundation to improve learning and increase the motivation of patients to learn and change. This motivation will be further strengthened by the use of the GlucoseMama monitoring system which will provide each patient with glucose tracking and individualized nutritional support.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gestational Diabetes
* Planning on delivering at home institution

Exclusion Criteria:

* Unwilling to participate.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of individuals requiring pharmacotherapy for treatment of gestational diabetes | 2 years

SECONDARY OUTCOMES:
Reduction in the number of neonates born large for gestational age. | 2 years
Increased number of individuals who are screened in the postpartum period for type 2 diabetes. | 2 years
Reduction in the number of infants with neonatal hypoglycemia. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States